CLINICAL TRIAL: NCT01087242
Title: Randomized，Double-blind，Dose Parallel Controlled, Multicentre Clinical Trail of Tang-min-Ling Pills and Placebo in Diabetes Mellitus(Liver-stomach Heat Retention Syndrome) (Phase Ⅲ)
Brief Title: Clinical Trail of Tang-min-Ling Pills in Type 2 Diabetes Mellitus
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Collaborators: Tianjin University of Traditional Chinese Medicine (Other); Liaoning University of Traditional Chinese Medicine (Other); Shanghai University of Traditional Chinese Medicine (Other); Beijing Hospital (Other Government); Tianjin Tasly Pharmaceutical Co., Ltd (Industry)
Responsible Party: Department of drug clinical trail institution, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2008L00307
Record Dates: First submitted 2010-03-09; First posted 2010-03-16 (Estimated); Last update posted 2010-03-16 (Estimated); Status verified 2009-05

CONDITIONS: Type 2 Diabetes
Keywords: Tang-min Lin pills; type 2 diabetes; liver and stomach heat retention; Evaluate the safety and efficacy of Tang-min Lin pills
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- controlled group (Placebo Comparator): Tang-min Lin analogue 6g,tid,po
  Interventions: Drug: Tang-min Lin pill
- Tang-min Lin pill (Experimental): Tang-min Lin pills 6g,tid,po
  Interventions: Drug: Tang-min Lin pill

INTERVENTIONS:
Drug: Tang-min Lin pill — Tang-min Lin pill 6g,tid,treat 12 weeks.

SUMMARY:
This is a randomized, doubled blind, dose-paralleled control, multi-centre clinical trail,to evaluate the efficacy of Tang-min-ling pills in the treatment of type 2 diabetes mellitus.

DETAILED DESCRIPTION:
Type 2 diabetes mellitus combined liver-stomach heat retension syndrome were recruited, which were divided into 3 groups .The patients were randomly taken with high-dosage (12g Tang-min-ling pills every time), low-dosage (6g Tang-min-ling pills every time), placebo by 3 times every day for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* initial treatment type 2 diabetic patient
* liver-stomach heat retention syndrome
* BMI ≥24kg/m2
* aged 30-65 years
* after screening stage(lifestyle intervention),Hba1C≥7.0%,FPG7.0-13.3mmol/L or PG2h>11.1mmol/L;
* voluntary signs the informed consent

Exclusion Criteria:

* have used anti-diabetes drug before more than 1 month
* used drug to control the blood sugar with 3 weeks
* diabetic ketosis,keto-acidosis,serious infection or trauma,major surgery within 1 month
* liver or kidney insufficiency,lung insufficiency,heart failure,acute myocardial infarction or other serious primary disease
* SBP/DBP >160mmHg/100 mmHg
* serious chronic diabetic complication
* chronic stomach-intestine disease,bad condition of the whole body
* pregnancy,preparing to pregnant,or breast-feed stage women
* allergic to TCM component
* mental disease
* allergic habitus
* attending to other clinical test
* attended this test before
* bibulosity and/or mental active drug,drug abuse or depend
* usually change the working environment,unstable live environment,etc.which will complied the inclusion
* unstable dose or type of anti-hypertension drug
* taking the drug or health food which will change the body weight

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2009-05; Primary Completion 2009-12 (Actual); Study Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
glycosylated hemoglobin | 0 and 12weeks after treatment

SECONDARY OUTCOMES:
fasting blood glucose,2-hour postprandial blood glucose,true insulin,TG,TG、LCL-C、HDL-C、BMI,waistline, hipline,TCM syndrome and sign | baseline and 12 week after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Wu S Tao, pro., Principal Investigator — Tian Jin university of tradtional chinese medicine; Lian F Mei, doctor, Study Chair — Guang'anmen Hospital of China Academy of Chinese Medical
Locations (4):
- China (4):
  - TCM school of Jiang Su province, Nanjing, Jiangsu
  - Liaoning University of Traditional Chinese Medicine, Shenyang, Liaoning
  - Shanghai University of Traditional Chinese Medicine, Shanghai, Shanghai Municipality
  - Tian Jin traditional chinese medicine university, Tianjin, Tianjin Municipality